CLINICAL TRIAL: NCT01982435
Title: Safety and Efficacy of Intravitreal Ranibizumab for Diabetic Macular Edema Previously Treated With Intravitreal Bevacizumab: A Randomized Dual Arm Comparative Dosing Trial
Brief Title: Safety and Efficacy of Ranibizumab for Diabetic Macular Edema
Acronym: REACT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Justis Ehlers (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Justis Ehlers, Staff physician / Sponsor-Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REACT Study
Record Dates: First submitted 2013-10-29; First posted 2013-11-13 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetes; Macular Edema
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I - Monthly (Other): Enrolled subjects will receive multiple open-label intravitreal injections of 0.3 mg ranibizumab administered every 28 days (+/- 7 days from the last treatment) for 12 months in the monthly group.
  Interventions: Drug: Ranibizumab
- Group II - Treat-and-Extend (Other): Enrolled subjects will initially receive 3 loading doses of open-label Ranibizumab 0.3 mg given via intravitreal injection every 28 days (+/- 7 days from the last treatment). After the third loading dose, the follow-up interval is determined by the Principal Investigator based on OCT results as stated in the protocol. The follow-up interval is increased by 2 weeks (+/- 7 days) at each visit up to a maximum interval of 12 weeks (+/- 7 days). There is criteria built into the protocol in case a reduction in the follow-up intervals becomes necessary based upon worsening OCT results.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Monthly injections of Intravitreal Ranibizumab 0.3 mg for 12 months in patients previously treated with Avastin for Diabetic Macular Edema.
  Other Names: Lucentis
  Arms: Group I - Monthly
Drug: Ranibizumab — Three Monthly injections of Intravitreal Ranibizumab 0.3 mg in patients previously treated with Avastin for Diabetic Macular Edema. Then follow-up visits may be extended by 2 weeks for a total of 12 months.
  Other Names: Lucentis
  Arms: Group II - Treat-and-Extend

SUMMARY:
The primary objective of the study is to assess the ocular and systemic adverse events of ranibizumab (Lucentis)for DME (diabetic macular edema) following previous treatment with intravitreal bevacizumab (Avastin).

DETAILED DESCRIPTION:
This is an open-label, Phase I/II study of intravitreally administered 0.3mg ranibizumab (Lucentis) in subjects with DME (diabetic macular edema) previously treated with intravitreal bevacizumab (Avastin) with a randomized comparative dosing strategy, monthly vs "treat-and-extend." Thirty patients total will be enrolled in the study, 15 in each group. This study will have a 1-year treatment period. The recruitment period will occur over 1 year with total potential study duration of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if the following criteria are met:

  * Ability to provide written informed consent and comply with study assessments for the full duration of the study
  * Age > 18 years
  * ETDRS best-corrected visual acuity of 20/25 to 20/320 in the study eye
  * Willing, committed, and able to return for ALL clinic visits and complete all study related procedures
  * At least 6 previous bevacizumab injections for diabetic macular edema in the last 12 months in the study eye.
  * At least 2 bevacizumab injections within 10 weeks and the most recent bevacizumab injection within 6 weeks of baseline study visits in the study eye.
  * Persistent foveal-involving diabetic macular edema based on presence of intraretinal and/or subretinal fluid by SDOCT in the foveal center at study entry in the study eye.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD (intrauterine device), or contraceptive hormone implant or patch.
* Intravitreal steroid or periocular steroid treatment within 3 months of study entry in the study eye.
* Focal/grid laser photocoagulation treatment within 3 months of study entry in the study eye.
* Panretinal photocoagulation treatment within 3 months of study entry in the study eye.
* Prior vitrectomy in the study eye
* History of retinal detachment in the study eye
* Prior trabeculectomy or other filtration surgery in the study eye
* Active intraocular inflammation in either eye
* Active ocular or periocular infection in either eye
* Active scleritis or episcleritis in either eye
* History of any other retinal vascular disease (e.g., retinal vein occlusion, retinal artery occlusion) in the study eye.
* Coexistent retinal disease other than diabetic retinopathy (e.g., AMD (age related macular degeneration), inherited retinal disease) in the study eye.
* Intraocular surgery within 3 months of study entry in the study eye.
* History of corneal transplant or corneal dystrophy in the study eye.
* Significant media opacities in study eye which may interfere with visual acuity in the study eye.
* Participation as a subject in any clinical study within 3 months of study entry.
* History of allergy to topical iodine
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justis Ehlers, M.D., Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cole Eye Institute, Cleveland Clinic, Cleveland, Ohio
  - Cole Eye Institute at Hillcrest Hospital, Mayfield Heights, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
Started | 15 | 12
Completed | 14 | 12
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (6.0) | 63.8 (6.4) | 63.1 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 5 | 6 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-severe Ocular Adverse Events
Description: As identified by eye examination (including visual acuity testing), identified by physical examination, subject reporting, and changes in vital signs. These outcome measures are also included in more detail in the adverse event section of the results.
Time Frame: 12 months
Population: Patients who exited the study early were accounted by using a last observation carried forward approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
Number analyzed (Participants) | 15 | 12
Participants
  Blurry Vision | 9 | 5
  Elevated IOP | 4 | 3
  Flashes | 3 | 3
  Vitreous Floaters | 3 | 2
  Dry eyes | 3 | 2
  Redness | 1 | 2
  Pruritus | 2 | 0
  Tearing | 1 | 1
  Non-severe ocular adverse events | 0 | 0
Statistical Analysis 1: Comparison: Group I - Monthly vs Group II - Treat-and-Extend; All analyses were performed with a significance level of 0.05 being assumed for all tests; Test type: Other — Measures were summarized using means, range and standard error of the means (SEM); p < 0.05, t-test, 2 sided — Two-sided paired t-tests and two-sided unpaired t-tests were respectively conducted to analyze efficacy endpoints between study initiation to end, and between monthly and TAE injection regimens

2. Primary Outcome: Number of Participants With Severe Ocular Adverse Events
Description: As identified by eye examination (including visual acuity testing), identified by physical examination, subject reporting, and changes in vital signs.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
Number analyzed (Participants) | 15 | 12
Participants
  Endophthalmitis | 0 | 0
  Retinal Detachment | 0 | 0

3. Primary Outcome: Number of Participants With Non-severe Non-ocular Adverse Event
Description: As identified by physical examination, subject reporting, and changes in vital signs. These outcome measures are also included in more detail in the adverse event section of the results.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
Number analyzed (Participants) | 15 | 12
Participants
  Blood and lymphatic adverse event | 1 | 0
  Cardiac adverse event | 8 | 4
  Gastrointestinal adverse event | 6 | 1
  General adverse event | 14 | 12
  Infectious advsere event | 1 | 0
  Metabolic adverse event | 3 | 2
  Musculoskeletal adverse event | 12 | 8
  Cyst, polyp and tumor adverse event | 3 | 0
  Nervous system adverse event | 2 | 0
  Psychiatric adverse event | 0 | 1
  Renal and urinary adverse event | 5 | 3
  Reproductive adverse event | 1 | 0
  Respiratory adverse event | 1 | 5
  Skin and subcutaneous adverse event | 8 | 2
  Vascular adverse event | 4 | 0

4. Primary Outcome: Number of Participants With Severe Non-ocular Adverse Event
Description: as for outcome 3
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
Number analyzed (Participants) | 15 | 12
Participants
  Hospitalizations | 6 | 3
  TIA | 1 | 0
  Stroke | 1 | 0

5. Secondary Outcome: Mean Change in BCVA
Description: Mean change in best-corrected visual acuity as assessed by the number of letters read correctly on the electronic ETDRS eye chart from baseline to months 6 and 12.
Time Frame: Months 6 and 12
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
Number analyzed (Participants) | 15 | 12
ETDRS letters
  Month 6 | .7 (8.1) | .7 (8.1)
  Month 12 | 2.1 (8.3) | 7.4 (10.4)

6. Secondary Outcome: Mean Change in Central Foveal Thickness
Description: Mean absolute change from baseline central foveal thickness at months 6 and 12 as measured by SDOCT (defined as the average thickness within the central 1 mm subfield)
Time Frame: Months 6 and 12
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
Number analyzed (Participants) | 15 | 12
microns
  Month 6 | -28.8 (173.4) | 104.1 (165.6)
  Month 12 | -80.9 (184.7) | -124 (157.6)

7. Secondary Outcome: Anatomically Dry Eyes by SDOCT
Description: Number of participants with an anatomically "dry" study eye by SDOCT at months 6 and 12
Time Frame: Months 6 and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
Number analyzed (Participants) | 15 | 12
Participants
  Month 6 | 0 | 0
  Month 12 | 0 | 1

8. Secondary Outcome: Gain in Vision Greater Than or Equal to 15 Letters
Description: Number of participants that gained greater than or equal to 15 letters of vision in their study eye at months 6 and 12.
Time Frame: Months 6 and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
Number analyzed (Participants) | 15 | 12
Participants
  Month 6 | 0 | 2
  Month 12 | 1 | 2

9. Secondary Outcome: Loss in Vision Greater Than or Equal to 15 Letters
Description: Number of participants that lost greater than or equal to 15 letters of vision in their study eye at months 6 and 12.
Time Frame: Months 6 and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
Number analyzed (Participants) | 15 | 12
Participants
  Month 6 | 1 | 0
  Month 12 | 1 | 0

10. Secondary Outcome: Participants With BCVA at 20/40 or Better
Description: Number of participants with 20/40 or better best-corrected visual acuity in their study eye at months 6 and 12.
Time Frame: Months 6 and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
Number analyzed (Participants) | 15 | 12
Participants
  Month 6 | 1 | 2
  Month 12 | 0 | 2

11. Secondary Outcome: Number of Participants With Angiographic Leakage
Description: Number of participants with angiographic leakage in their study eye measured from baseline to months 3, 6 and 12 (i.e. presence of leakage).
Time Frame: 3, 6 and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
Number analyzed (Participants) | 15 | 12
Participants
  3 month | 15 | 12
  6 month | 15 | 12
  12 month | 15 | 12

12. Secondary Outcome: Number of Participants With Nonperfusion
Description: Number of participants with peripheral nonperfusion in their study eye from baseline to months 3, 6, and 12 (i.e. presence of ischemia).
Time Frame: 3, 6 and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
Number analyzed (Participants) | 15 | 12
Participants
  3 months | 13 | 9
  6 months | 13 | 10
  12 months | 12 | 9

ADVERSE EVENTS:
Arm/Group | Group I - Monthly | Group II - Treat-and-Extend
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/12
Serious Adverse Events (participants affected / at risk) | 6/15 | 3/12
Other Adverse Events (participants affected / at risk) | 15/15 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I - Monthly (N=15) | Group II - Treat-and-Extend (N=12)
Worsening of Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0)
POSSIBLE CELLULITIS TO RIGHT LOWER EXTREMITY (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHEMIC ATTACK (Cardiac disorders) | 1 (1) | 0 (0)
ACUTE INFARCT STROKE (Cardiac disorders) | 1 (1) | 0 (0)
UNSTABLE ANGINA AND CHEST PAIN (Cardiac disorders) | 1 (1) | 0 (0)
VERTIGO (General disorders) | 0 (0) | 1 (1)
LARGE OVARIAN NEOPLASM (Reproductive system and breast disorders) | 1 (1) | 0 (0)
HOSPITALIZED FOR PERITONITIS (Renal and urinary disorders) | 1 (1) | 0 (0)
HOSPITALIZED FOR ANGINA/SOB (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HOSPITALIZED FOR DIABETIC RIGHT HEEL ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HOSPITALIZED FORCONFUSION/SLURRED SPEECH AFTER FALL (Social circumstances) | 1 (1) | 0 (0)
HOSPITALIZED FOR RECURRENT SOB, LEG EDEMA (General disorders) | 1 (1) | 0 (0)
HOSPITALIZATION FOR GANGRENE (Infections and infestations) | 1 (1) | 0 (0)
HOSPITALIZATION R DIABETIC FOOT ULCER INFECTION (Infections and infestations) | 1 (1) | 0 (0)
HOSPITALIZATION FOR TOTAL HYSTERECTOMY (Reproductive system and breast disorders) | 0 (0) | 1 (1)
HOSPITALIZATION FOR HYPERKALEMIA (Endocrine disorders) | 0 (0) | 1 (1)
HOSPITALIZATION FOR GANGRENE/AMPUTATION (Infections and infestations) | 1 (1) | 0 (0)
HOSPITALIZATION FOR OSTEOMYELITIS/AMPUTATION (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I - Monthly (N=15) | Group II - Treat-and-Extend (N=12)
Decreased Vision (Eye disorders) | 5 (5) | 4 (4)
Hypertension (Cardiac disorders) | 4 (4) | 2 (2)
Flu-like symptoms (General disorders) | 4 (4) | 5 (5)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Difficulty with reading (Eye disorders) | 5 (5) | 5 (5)
Difficulty with driving (General disorders) | 2 (2) | 2 (2)
Hyperglycemic episode (General disorders) | 0 (0) | 1 (1)
Edema (Vascular disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Worsening of diabetes (Renal and urinary disorders) | 3 (4) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Weight gain (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Foreign Body Sensation (Eye disorders) | 2 (2) | 1 (1)
Hypoglycemic episode (General disorders) | 2 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Stye (Eye disorders) | 3 (3) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Urinary Tract infection (Renal and urinary disorders) | 2 (3) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain from fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Chest pain (Cardiac disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Generalized rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Headache (General disorders) | 2 (2) | 1 (1)
Thyroid cancer (General disorders) | 1 (1) | 0 (0)
Uterine cancer suspect (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bladder cancer (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Epiretinal Membrane (Eye disorders) | 0 (0) | 3 (3)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Vitamin Deficiency (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Elevated microalbumin (General disorders) | 0 (0) | 1 (1)
Ocular irritation (Eye disorders) | 6 (6) | 2 (2)
Eye Discharge (Eye disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Generalized weakness (General disorders) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (General disorders) | 1 (1) | 0 (0)
Benign polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Thalassemia Trait (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Optic neuropathy (Eye disorders) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Atherosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elevated Creatinine levels (General disorders) | 0 (0) | 1 (1)
Sun damage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Elevated d-Dimer (General disorders) | 1 (1) | 0 (0)
Hypomagnesemia (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thyroid nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OSA Worsening (General disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 0 (0) | 1 (1)
Worsening of cataracts (Eye disorders) | 2 (2) | 0 (0)
Cold Sore (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperlipidemia (General disorders) | 1 (1) | 0 (0)
Glare in vision (Eye disorders) | 2 (2) | 0 (0)
Elevated INR (General disorders) | 0 (0) | 1 (1)
Pruritus after fluorescein dye (General disorders) | 0 (0) | 1 (1)
Asymptomatic Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bullous eruption on glans (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus on neck (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Insomnia - worsening (General disorders) | 0 (0) | 1 (1)
Posterior Vitreous Detachment (Eye disorders) | 0 (0) | 1 (1)
Hyperkalemia (General disorders) | 0 (0) | 1 (1)
Ptosis (Eye disorders) | 0 (0) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ocular swelling (Eye disorders) | 0 (0) | 1 (1)
Medicamentosa suspect (General disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (3) | 0 (0)
Chronic angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Lower extremity sprain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Subconjunctival Hemorrhage (Eye disorders) | 2 (2) | 1 (1)
Tingling sensation in feet (General disorders) | 1 (1) | 0 (0)
Puncture wound (Eye disorders) | 1 (1) | 0 (0)
Elevated Heart Rate (Cardiac disorders) | 1 (2) | 0 (0)
Elevated FBS (General disorders) | 1 (1) | 0 (0)
Staph infection of wound on ankle (Infections and infestations) | 1 (1) | 0 (0)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Difficulty with watching television (Eye disorders) | 1 (1) | 3 (3)
Addison's Disease worsening (General disorders) | 1 (1) | 0 (0)
Worsening of trigger finger (General disorders) | 1 (1) | 0 (0)
Elevated TSH levels (General disorders) | 1 (1) | 0 (0)
SOB episode - allergy to Zanaflex (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The relatively small sample size of eyes and short 1 year duration makes it challenging to extrapolate data to generate clinical management guidelines. The lack of a control group is an important limitation to recognize that also limits conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT01982435/Prot_000.pdf
  • Statistical Analysis Plan (2013-11-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT01982435/SAP_002.pdf